CLINICAL TRIAL: NCT06149221
Title: Using Direct Non-thermal Atmospheric Pressure Plasma With Penetration Enhancement for the Treatment of Hair Loss
Brief Title: Penetration-enhanced Direct DBD Non-thermal Plasma for Hair Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Peter C. Friedman (Industry)
Responsible Party: Sponsor-Investigator, Dr. Peter C. Friedman, President, The Skin Center Dermatology Group
Organization: The Skin Center Dermatology Group (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCAP
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Androgenetic Alopecia
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NTAP treatment (Experimental): Treatment arm subjects receive the trial intervention
  Interventions: Device: NTAP

INTERVENTIONS:
Device: NTAP — Cold plasma is generated and applied to the scalp area, which was previously soaked with normal saline

SUMMARY:
In-office applied non-thermal atmospheric pressure plasma treatment on NS pretreated scalp

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild-to moderate androgenetic alopecia
* ability to keep in-person follow-up appointments

Exclusion Criteria:

* any inflammatory scalp condition
* starting or discontinuing any hair loss treatments within 6 months of start date
* allergy to any components of the carrier solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-12 (Actual); Study Completion 2024-04-12 (Actual)

PRIMARY OUTCOMES:
Presence of detectable hair growth | 3 months and 6 months
  Presence of hair growth as measured using the HairMetrix device

SECONDARY OUTCOMES:
Adverse effects related to the treatment | throughout study completeion, 6 months
  Patients are monitored for adverse effects, including but not limited to irritation, itch, inflammation, scaling, redness, rash, peeling, blistering

CONTACTS AND LOCATIONS:
Locations (1):
- The Skin Center Dermatology Group, New City, New York, United States

IPD SHARING:
Plan to Share IPD: No